CLINICAL TRIAL: NCT01842035
Title: Heart Rate Response to Regadenoson and Sudden Cardiac Death
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Astellas Scientific & Medical Affairs, Inc. (Industry)
Responsible Party: Principal Investigator, Fadi Hage, MD, MD, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REGA 12D05
Record Dates: First submitted 2013-03-13; First posted 2013-04-29 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Left Ventricular Systolic Dysfunction; Sudden Cardiac Death
Keywords: Implantable cardiac defibrillator; regadenoson; sudden cardiac death; heart rate response
MeSH Terms: conditions — Ventricular Dysfunction, Left; Death, Sudden, Cardiac | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regadenoson (Experimental): Prior to the implantation of a clinically indicated ICD, the heart rate response to regadenoson will be assessed. Regadenoson will be administered intravenously as a fixed intravenous bolus dose of 400 μg followed by a 5 mL saline flush. Medications (including beta-blockers) will be withheld on the morning of the test. The heart rate and blood pressure will be measured at baseline and every minute after regadenoson bolus for at least 5 minutes and until the heart rate and blood pressure are clearly returning towards baseline.
  --------------------------------------------------------------------------------
  Interventions: Drug: regadenoson

INTERVENTIONS:
Drug: regadenoson — Prior to the implantation of a clinically indicated ICD, the heart rate response to regadenoson will be assessed. Regadenoson will be administered intravenously as a fixed intravenous bolus dose of 400 μg followed by a 5 mL saline flush. Medications (including beta-blockers) will be withheld on the morning of the test. The heart rate and blood pressure will be measured at baseline and every minute after regadenoson bolus for at least 5 minutes and until the heart rate and blood pressure are clearly returning towards baseline.
  Other Names: Lexiscan

SUMMARY:
The purpose of this study is to determine whether a blunted heart rate response to regadenoson is an independent predictor of sudden cardiac death.

DETAILED DESCRIPTION:
In patients with heart failure and in those with a history of sudden cardiac death, an Implantable Cardiac Defibrillator (ICD) reduces death rates. However, not all patients with an ICD receive appropriate therapy from it. Inappropriate ICD shocks are common and are associated with worse quality of life and increased death rate. We hope to establish a better predictor of risk of sudden cardiac death and of response to ICD. We are conducting a prospective observational study of 150 patients (18-80 years) with an indication for ICD implantation for primary prevention of sudden cardiac death. Prior to the implantation of a clinically indicated ICD, the heart rate response to regadenoson will be assessed. Regadenoson will be administered intravenously as a fixed intravenous bolus dose of 400 μg followed by a 5 mL saline flush.

The main objectives of this proposal are to investigate whether:

1. A blunted heart rate response to regadenoson is an independent predictor of sudden cardiac death.
2. A blunted heart rate response to regadenoson can be used as a predictor of response to ICD on top of traditionally used indicators.

We Hypothesize that:

1. Patients with a blunted heart rate response to regadenoson are at higher risk of sudden cardiac death (death or appropriate cardiac defibrillation). This risk is maintained after controlling for age, gender, left ventricular ejection fraction, heart failure symptoms and medication use.
2. Patients with a normal heart rate response to regadenoson have a low rate of events (death or appropriate cardiac defibrillation) despite meeting current indications for having an ICD.

ELIGIBILITY:
Inclusion criteria:

* Age 19-80 years
* Female subjects must be (a) at least one year post-menopause or surgically sterile or (b) be non-pregnant and (c) non-lactating.
* Subject must be able and willing to provide written informed consent
* Subject must be referred for a clinically indicated ICD and fall into one of the following groups:

  * subjects with left ventricular ejection fraction less than 35% due to prior myocardial infarction who are at least 40 days post-myocardial infarction and are in NYHA functional Class II or III.
  * subjects with non-ischemic dilated cardiomyopathy who have a left ventricular ejection fraction less than or equal to 35% and who are in NYHA functional Class II or III.
  * Subjects with left ventricular dysfunction due to prior myocardial infarction who are at least 40 days post-myocardial infarction, have a left ventricular ejection fraction less than 30%, and are in NYHA functional Class I.

Exclusion Criteria:

* Female subject who is pregnant or lactating
* Subject with active severe asthma or chronic obstructive pulmonary disease which, in the Investigator's opinion, places the subject at risk for severe bronchoconstriction
* Treatment with dipyridamole, theophylline, aminophylline or pentoxifylline within 24 hours of receiving regadenoson
* Treatment with any investigational drug within 30 days or 5 half lives - whichever is longer prior to study entry
* Subject with any prior allergic response to aminophylline or other contraindication to receiving intravenous regadenoson
* Subjects with second or third degree atrioventricular block or dependent on pacemaker
* Subject with uncontrolled severe hypertension (systolic > 200 mmHg or diastolic >120 mmHg) or pretreatment hypotension (systolic BP <90 mmHg)
* Subject with hemodynamically significant aortic stenosis or outflow tract obstruction
* Subject with decompensated heart failure (NYHA functional class IV)
* Subject with acute myocardial infarction, new onset of ischemia, percutaneous coronary intervention, or coronary artery bypass grafting within 30 days of receiving regadenoson
* Subject is on dialysis for end stage renal disease or has an estimated glomerular filtration rate < 15 mL/min
* Subjects with cardiac transplantation

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fadi G Hage, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

REFERENCES:
- [Background] Hage FG, Heo J, Franks B, Belardinelli L, Blackburn B, Wang W, Iskandrian AE. Differences in heart rate response to adenosine and regadenoson in patients with and without diabetes mellitus. Am Heart J. 2009 Apr;157(4):771-6. doi: 10.1016/j.ahj.2009.01.011. Epub 2009 Mar 6. PMID 19332209
- [Background] Hage FG, Perry G, Heo J, Iskandrian AE. Blunting of the heart rate response to adenosine and regadenoson in relation to hyperglycemia and the metabolic syndrome. Am J Cardiol. 2010 Mar 15;105(6):839-43. doi: 10.1016/j.amjcard.2009.11.042. PMID 20211328
- [Background] Hage FG, Dean P, Bhatia V, Iqbal F, Heo J, Iskandrian AE. The prognostic value of the heart rate response to adenosine in relation to diabetes mellitus and chronic kidney disease. Am Heart J. 2011 Aug;162(2):356-62. doi: 10.1016/j.ahj.2011.05.014. Epub 2011 Jul 18. PMID 21835298
- [Background] Hage FG, Dean P, Iqbal F, Heo J, Iskandrian AE. A blunted heart rate response to regadenoson is an independent prognostic indicator in patients undergoing myocardial perfusion imaging. J Nucl Cardiol. 2011 Dec;18(6):1086-94. doi: 10.1007/s12350-011-9429-1. Epub 2011 Jul 22. PMID 21785922
- [Background] Iqbal FM, Al Jaroudi W, Sanam K, Sweeney A, Heo J, Iskandrian AE, Hage FG. Reclassification of cardiovascular risk in patients with normal myocardial perfusion imaging using heart rate response to vasodilator stress. Am J Cardiol. 2013 Jan 15;111(2):190-5. doi: 10.1016/j.amjcard.2012.09.013. Epub 2012 Oct 27. PMID 23111139

RESULTS

PARTICIPANT FLOW:
Groups:
- Regadenoson: Prior to the implantation of a clinically indicated ICD, the heart rate response to regadenoson will be assessed. Regadenoson will be administered intravenously as a fixed intravenous bolus dose of 400 μg followed by a 5 mL saline flush. Medications (including beta-blockers) will be withheld on the morning of the test. The heart rate and blood pressure will be measured at baseline and every minute after regadenoson bolus for at least 5 minutes and until the heart rate and blood pressure are clearly returning towards baseline.
  --------------------------------------------------------------------------------
  regadenoson: Prior to the implantation of a clinically indicated ICD, the heart rate response to regadenoson will be assessed. Regadenoson will be administered intravenously as a fixed intravenous bolus dose of 400 μg followed by a 5 mL saline flush. Medications (including beta-blockers) will be withheld on the morning of the test. The heart rate and blood pressure will be measured at baseline and every minute after regadenoson bolus for at least 5 minutes and until the heart rate and blood pressure are clearly returning towards baseline.
Period: Overall Study
Arm/Group | Regadenoson
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Regadenoson
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] — Age: mean and standard deviation
  years | 60 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 36
  White | 54
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Sudden Cardiac Death
Description: Sudden cardiac death will be defined as death within 1 hour of symptom onset, or an unobserved death in which the patient was seen and known to be doing well within 24 hours of death. Survivors of aborted sudden cardiac death, resuscitated cardiac arrest, and those receiving appropriate ICD therapy will also be considered to have experienced sudden cardiac death and will be included in the primary end point.
Time Frame: Until end of follow-up, median follow-up 40 months
Measure: Count of Participants; unit: Participants
Groups:
- Heart Rate Response Greater Than Median: Heart rate response >= 24%
- Heart Rate Response Less Than Median: Heart rate response < 24%
Arm/Group | Heart Rate Response Greater Than Median | Heart Rate Response Less Than Median
Number analyzed (Participants) | 44 | 46
Participants | 2 | 6

2. Secondary Outcome: All-cause Death
Description: death from any cause
Time Frame: Until end of follow-up, median follow-up 40 months
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Rate Response Greater Than Median | Heart Rate Response Less Than Median
Number analyzed (Participants) | 44 | 46
Participants | 8 | 8

3. Secondary Outcome: First Appropriate ICD Therapy
Description: antitachycardia pacing therapy or shock for tachyarrhythmia determined by evaluation of the clinical information and by device diagnostics to be either ventricular fibrillation or ventricular tachycardia
Time Frame: Until end of follow-up, median follow-up 40 months
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Rate Response Greater Than Median | Heart Rate Response Less Than Median
Number analyzed (Participants) | 44 | 46
Participants | 6 | 12

4. Secondary Outcome: Inappropriate ICD Therapy
Description: unnecessary antitachycardia pacing or shock delivered by the ICD for a rhythm that is not a true ventricular fibrillation or ventricular tachycardia
Time Frame: Until end of follow-up, median follow-up 40 months
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Rate Response Greater Than Median | Heart Rate Response Less Than Median
Number analyzed (Participants) | 44 | 46
Participants | 3 | 2

5. Secondary Outcome: All-cause Death or First Appropriate ICD Therapy
Description: death or antitachycardia pacing therapy or shock for tachyarrhythmia determined by evaluation of the clinical information and by device diagnostics to be either ventricular fibrillation or ventricular tachycardia
Time Frame: Until end of follow-up, median follow-up 40 months
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Rate Response Greater Than Median | Heart Rate Response Less Than Median
Number analyzed (Participants) | 44 | 46
Participants | 13 | 16

6. Secondary Outcome: Sudden Cardiac Death or Appropriate ICD Therapy
Description: Sudden cardiac death or antitachycardia pacing therapy or shock for tachyarrhythmia determined by evaluation of the clinical information and by device diagnostics to be either ventricular fibrillation or ventricular tachycardia
Time Frame: Until end of follow-up, median follow-up 40 months
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Rate Response Greater Than Median | Heart Rate Response Less Than Median
Number analyzed (Participants) | 44 | 46
Participants | 8 | 15

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored for 1 day and deaths were monitored until end of follow-up, median of 40 months
Description: Adverse events were monitored for 1 day while outcomes were monitored until end of follow-up.
Arm/Group | Regadenoson
All-Cause Mortality (participants affected / at risk) | 16/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 24/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regadenoson (N=90)
symptomatic hypotension (Vascular disorders) | 0 (0)
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0)
flushing (Skin and subcutaneous tissue disorders) | 11 (11)
chest pain (Cardiac disorders) | 1
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Gastrointestinal symptoms (Gastrointestinal disorders) | 9 (9)
Ventricular tachycardia (Cardiac disorders) | 0 (0)

LIMITATIONS AND CAVEATS:
The lower than planned sample size decreased the power of the study. To partially compensate, we allowed for longer than planned follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT01842035/Prot_SAP_000.pdf